CLINICAL TRIAL: NCT06342375
Title: Enrollment Barriers, Procedural Denials, and Loss of Medicaid Coverage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Covering Wisconsin (Unknown); Arnold Ventures (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-0434; A538500 (Other: UW- Madison); Protocol Version 4/17/2025 (Other: UW- Madison); SMPH/POP HEALTH SCI/POP HLTH (Other: UW- Madison)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-04

CONDITIONS: No Medicaid Coverage
Keywords: Medicaid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Outreach (Experimental): People in this cohort will receive a live outbound call from a Navigator
  Interventions: Other: Outbound phone call
- Pre-recorded Outreach (Experimental): People in this cohort will receive a pre-recorded outbound call providing a hotline number
  Interventions: Other: Outbound phone call
- No outreach (No Intervention): People in this cohort will not receive outreach of any kind

INTERVENTIONS:
Other: Outbound phone call — Participants will receive either a live or pre-recorded outbound phone call
  Arms: Live Outreach; Pre-recorded Outreach

SUMMARY:
The goal of this study is to try new outreach methods to improve access to Medicaid for those who lost Medicaid for procedural reasons. The main questions it aims to answer are:

1. How does a live phone call from a Navigator impact Medicaid enrollment among people who lost Medicaid coverage for procedural reasons?
2. What is the effectiveness of outreach using a live call rather than a pre-recorded call?

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Medicaid
* Lost Medicaid coverage between June 2024 and November 2025

Exclusion Criteria:

* Preferring a language other than English, Spanish, or Hmong
* No working phone number

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425000 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of people who successfully renew their Medicaid coverage within 3 months of receiving the live outbound call | 3 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.

SECONDARY OUTCOMES:
Duration of coverage gaps | 6 months
  Duration of gaps will be measured using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.
Number of people who successfully renew their Medicaid coverage within 6 months of receiving the live outbound call | 6 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.
Number of people who successfully renew their Medicaid coverage within 6 months of receiving the pre-recorded outbound call | 6 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Myerson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No